CLINICAL TRIAL: NCT06594913
Title: Eating Disorders Genetics Initiative 2
Acronym: EDGI2
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Queensland Institute of Medical Research (Other); Karolinska Institutet (Other); National Institute of Mental Health (NIMH) (NIH); University of Otago (Other); University of Aarhus (Other); Yale University (Other); Comenzar de Nuevo, AC (Other); University of Sydney (Other)
Responsible Party: Sponsor
Other Study IDs: 23-2887; R01MH136149 (NIH); R01MH136157 (NIH); R01MH136156 (NIH)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Avoidant Restrictive Food Intake Disorder
Keywords: severe and enduring eating disorder; genetics; mental health; disordered eating; environmental factors
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Avoidant Restrictive Food Intake Disorder; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Saliva samples will be collected for DNA extraction. Both saliva samples and DNA will be retained in biorepositories.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Anorexia nervosa: Individuals with a self-reported lifetime history of anorexia nervosa.
  Interventions: Other: Eating disorder diagnosis group
- Bulimia nervosa: Individuals with a self-reported lifetime history of bulimia nervosa.
  Interventions: Other: Eating disorder diagnosis group
- Binge-eating disorder: Individuals with a self-reported lifetime history of binge-eating disorder.
  Interventions: Other: Eating disorder diagnosis group
- ARFID: Individuals with a self-reported lifetime history of avoidant restrictive food intake disorder.
  Interventions: Other: Eating disorder diagnosis group
- Control: Individuals with no history of disordered eating behaviors or symptoms
  Interventions: Other: Eating disorder diagnosis group

INTERVENTIONS:
Other: Eating disorder diagnosis group — This is an observational study, no active intervention is applied. Participants are assigned to an eating disorder diagnosis group based on their lifetime history of disordered eating behaviors and symptoms.

SUMMARY:
The overarching intention of the Eating Disorder Genetics Initiative 2 (EDGI2) is to increase sample size, diversity, and eating disorder phenotypes. The investigators are enrolling 20,000 new participants with anorexia nervosa (AN), bulimia nervosa (BN), binge-eating disorder (BED), avoidant/restrictive food intake disorder (ARFID), and controls in the US, Mexico, Australia, New Zealand, Sweden, and Denmark. A primary study goal is to enroll at least 30% of participants from underrepresented groups. Participants are asked to complete a series of questionnaires and submit a saliva sample for genotyping. The goal is to better understand eating disorders and how they relate to each other so that better treatments can be developed.

ELIGIBILITY:
Inclusion Criteria:

* A lifetime history of anorexia nervosa, bulimia nervosa, binge-eating disorder, avoidant restrictive food intake disorders or no history of any disordered eating behavior, based on DSM-5 criteria algorithms
* Age 12-99 years, depending on country. (US enrollment age is 18-99)

Exclusion Criteria:

* History of subthreshold disordered eating behaviors.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Interested individuals from the United States, Mexico, Australia, New Zealand, and Sweden who meet criteria may participate within their respective country.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Identified with an Eating Disorder Diagnosis by Category | Baseline
  The ED100Kv4 is a web-based diagnostic questionnaire, based on the Structured Clinical Interview for Axis 1 Disorders, that applies algorithms to participant responses. The number of participants with each diagnosis (AN, BN, BED, ARFID, and control) will be reported.
Age of eating disorder onset | Baseline
  Age of eating disorder onset will be considered as the age of first eating disorder symptom as self-reported in the ED100Kv4 questionnaire (ED100K). Age of onset will be reported for each eating disorder group.

SECONDARY OUTCOMES:
Current Disordered Eating Symptoms | Baseline
  Current eating disorder symptoms will be determined by self-report responses on the Eating Disorder Examination Questionnaire (EDEQ), the Binge Eating Disorder Screener-(BEDS7), the Nine Item ARFID Screen (NIAS), Muscle Dysmorphic Disorder Inventory (MDDI), the Drive for Muscularity Scale (DMS), and food insecurity. Items in all assessments ask about current symptoms related to eating disorders. The assessments sum scores to create subscales where higher scores indicate more eating disorder pathology and the scores taken together reveal the current disordered eating status of participants. Subscale sores will be reported for the total sample.
Mental Health and Behavior | Baseline
  Current mental health symptoms (depression, anxiety, obsessive-compulsive disorder, autism, and attention-deficit/hyperactivity disorder [ADHD]) are assessed using the Patient Health Questionnaire (PHQ), Generalized Anxiety Disorder 7 (GAD7), Obsessional Compulsive Inventory - Revised (OCI-R), Autism Spectrum Quotient (AQ10), and Adult ADHD Self-Report Scale (ASRS).The assessments sum scores to create subscales where higher scores indicate more mental health symptoms and the scores taken together provide insight to current comorbidity of participants. Subscale sores will be reported for the entire sample
Mood - Lifetime history of mood and anxiety disorders | Baseline
  The GLAD questionnaire asks about lifetime history of mood and anxiety symptoms. Algorithms based on Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) criteria will be applied to data to report lifetime history of mood and anxiety disorders.
Self-Violence | Baseline
  A series of questions will be asked about suicidality and self-harm. The number and percent of participants indicating suicidality and self-harm will be reported.
Lifetime Substance Use | Baseline
  Adapted to lifetime use, Alcohol Use Disorders Identification Test (AUDIT; 10 times) and the Drug Use Disorders Identification Test (DUDIT) are administered along with the heaviness of smoking and and questions about vaping. The AUDIT, DUDIT, and heaviness of smoking are scored using published algorithms. The prevalence of lifetime substance use will be reported for each eating disorder group.
Life-Events | Baseline
  A modified version of Life Events Checklist for DSM-5 (LEC-5) is administered to collect information about 20 adverse events experienced, the age those events were first experienced, and the degree of trauma that resulted from the life events. The number and percent of each life event experienced will be reported for each eating disorder group.
Eating Disorder Quality of Life | Baseline
  Eating disorder quality of life is measured with the Eating Disorder Quality of Life (EDQL) self-report questionnaire. The EDQL asks 25 items about the psychological, physical, financial, and work/school impact of an eating disorder over the past 30 days. Items are scored never (0), rarely (1), sometimes (2), often (3), or always (4). Items are summed for a total score ranging from 0-100, representing the overall impact of an eating disorder on life quality. Higher scores indicate a more significant impact of the eating disorder on life quality. Scores will be reported for each eating disorder group.
Compulsive Exercise Test | Baseline
  Maladaptive exercise is evaluated using the Compulsive Exercise Test. A total of 24 questions ask about excessive or problematic exercise. Response options are on a 6-point Likert scale. There are 5 subscales, which are scored according to published criteria. Higher scores indicate greater pathology. Scores will be reported for each eating disorder group.
Perfectionism | Baseline
  A shortened version (12 items) of the Multidimensional Perfectionism Scale (MPS) is used to assess 3 features of perfectionism: doubts about actions, concern over mistakes, and personal standards. Response options are on a 5-point Likert scale. Greater scores indicate higher perfectionism. Scores will be reported for each eating disorder group.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Bulik, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States
- QIMR Berghofer, Brisbane, Queensland, Australia
- Comenzar de Nuevo, Monterrey, Mexico
- University of Otago, Christchurch, Canterbury, New Zealand
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and scripts will be made available to the general scientific community at the conclusion of the investigation. Specifically, phenotype data from the United States, Mexico, Australia, and New Zealand will be submitted to the database of Genotypes and Phenotypes (dbGaP) and National Institute of Mental Health Repository & Genetics Resource (NRGR) and genotype data to dbGaP. Data from Sweden will be made available on the Federated European Genome-phenome Archive.
Supporting Information: Study Protocol, ICF
Time Frame: Assessment phenotype data will be submitted within 6 months after the end of the study. Genotype data will be submitted after the first set of analyses with these data are complete. All data will be available as long as the repositories maintain the datasets (indefinitely).
Access Criteria: The databases are controlled-access meaning that individuals who wish to have access to the data must apply to the respective repository and meet all of their criteria.
URL: https://nda.nih.gov/nda/access-data-info.html

REFERENCES:
- [Derived] Berthold N, MacDermod CM, Thornton LM, Parker R, Morales SAC, Hog L, Kennedy HL, Guintivano J, Sullivan PF, Crowley JJ, Johnson JS, Birgegard A, Fundin BT, Frans E, Xu J, Ngati Pukenga MP, Miller AL, Aguilar MV, Barakat S, Abdulkadir M, White JP, Larsen JT, Trujillo E, Winterman B, Zhang R, Lawson R, Wonderlich S, Wonderlich J, Schaefer LM, Mehler PS, Oakes J, Foster M, Gaudiani J, Vacuan ETC, Compte EJ, Petersen LV, Yilmaz Z, Micali N, Jordan J, Kennedy MA, Maguire S, Huckins LM, Lu Y, Dinkler L, Martin NG, Bulik CM. The Eating Disorders Genetics Initiative 2 (EDGI2): study protocol. BMC Psychiatry. 2025 May 26;25(1):532. doi: 10.1186/s12888-025-06777-5. PMID 40419993